CLINICAL TRIAL: NCT02023879
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Evaluating the Efficacy and Safety of Alirocumab in Patients With Primary Hypercholesterolemia Not Treated With a Statin
Brief Title: Phase III Study To Evaluate Alirocumab in Patients With Hypercholesterolemia Not Treated With a Statin (ODYSSEY CHOICE II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC13786; 2013-002659-14 (EudraCT Number); U1111-1146-3517 (Other: UTN)
Record Dates: First submitted 2013-12-06; First posted 2013-12-30 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Diet

STUDY DESIGN:
Intervention Model Description: A double-blind treatment period of 24 weeks (3 parallel arms) followed by an open-label extension period (single arm)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking during the double-blind treatment period
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Q2W (Placebo Comparator): Period 1: Placebo (for Alirocumab) subcutaneous (SC) injection every 2 weeks (Q2W) added to stable non-statin lipid modifying therapy (LMT) or diet alone for 24 weeks.
  Period 2: Alirocumab 150 mg SC injection every 4 weeks (Q4W) from Week 24 until second quarter 2017 or until the drug is commercially available in the country, whatever occurred first. Alirocumab dose could be either up-titrated to 150 mg Q2W from Week 36 or maintained according to the investigator judgement and low-density lipoprotein cholesterol (LDL-C) values. Subsequent down titration to 150 mg Q4W was allowed.
  Interventions: Drug: Alirocumab; Drug: Placebo (for Alirocumab); Drug: Non-statin LMT; Other: Diet Alone
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W (Calibrator) (Other): Period 1: Alirocumab 75 mg SC injection Q2W added to stable non-statin LMT or diet alone for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when targeted LDL-C levels at Week 8 were not achieved i.e. LDL-C ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) depending on cardiovascular risk or <30% LDL-C reduction from baseline.
  Period 2: Alirocumab 150 mg SC injection Q4W from Week 24 until second quarter 2017 or until the drug is commercially available in the country, whatever occurred first. Alirocumab dose could be either up-titrated to 150 mg Q2W from Week 36 or maintained according to the investigator judgement and LDL-C values. Subsequent down titration to 150 mg Q4W was allowed.
  Interventions: Drug: Alirocumab; Drug: Non-statin LMT; Other: Diet Alone
- Alirocumab 150 mg Q4W/Up to 150 mg Q2W (Experimental): Period 1: Alirocumab 150 mg SC injection Q4W alternating with placebo (for alirocumab) Q4W added to stable non-statin LMT or diet alone for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when targeted LDL-C levels at Week 8 were not achieved i.e. LDL-C ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) depending on cardiovascular risk or <30% LDL-C reduction from baseline.
  Period 2: Alirocumab 150 mg SC injection Q4W from Week 24 until second quarter 2017 or until the drug is commercially available in the country, whatever occurred first. Alirocumab dose could be either up-titrated to 150 mg Q2W from Week 36 or maintained according to the investigator judgement and LDL-C values. Subsequent down titration to 150 mg Q4W was allowed.
  Interventions: Drug: Alirocumab; Drug: Placebo (for Alirocumab); Drug: Non-statin LMT; Other: Diet Alone

INTERVENTIONS:
Drug: Alirocumab — Solution for injection in the abdomen, thigh, or outer area of the upper arm by self-injection or by another designated person using auto-injector (also known as pre-filled pen).
  Other Names: SAR236553; REGN727; Praluent®
Drug: Placebo (for Alirocumab) — Solution for injection in the abdomen, thigh, or outer area of the upper arm by self-injection or by another designated person using auto-injector (also known as pre-filled pen).
  Arms: Alirocumab 150 mg Q4W/Up to 150 mg Q2W; Placebo Q2W
Drug: Non-statin LMT — Ezetimibe or Fenofibrate at stable dose as background therapy.
Other: Diet Alone — Stable cholesterol-lowering diet as background therapy.

SUMMARY:
Primary Objective:

To demonstrate the reduction of low-density lipoprotein cholesterol (LDL-C) by a regimen of Alirocumab including a starting dose of 150 mg every 4 weeks (Q4W) as add-on to non-statin lipid modifying background therapy or as monotherapy in comparison with placebo in participants with primary hypercholesterolemia not treated with a statin.

Secondary Objective:

* To evaluate the effects on other lipid parameters of Alirocumab 150 mg Q4W versus placebo.
* To evaluate the safety and tolerability of Alirocumab 150 mg Q4W.

Alirocumab 75 mg Q2W was added as a calibrator arm.

DETAILED DESCRIPTION:
The core study duration was approximately 35 weeks per participant (screening: 3 weeks, double-blind treatment period: 24 weeks; follow-up: 8 weeks). Participants who successfully completed the treatment period had the possibility to participate in an optional open-label treatment period with Alirocumab 150 mg Q4W until second quarter 2017 or until the drug is commercially available in the country, whatever occurred first.

ELIGIBILITY:
Inclusion criteria:

Participants with primary hypercholesterolemia (heterozygous familial hypercholesterolemia [heFH] or non-FH) not adequately controlled with their non-statin LMT (either ezetimibe or fenofibrate) or diet alone.

Exclusion criteria:

* LDL-C <70 mg/dL (1.81 mmol/L) at screening for statin intolerant participants at very high cardiovascular (CV) risk;
* LDL-C <100 mg/dL (<2.59 mmol/L) at screening for statin intolerant participants at high or moderate CV risk or, participants not fulfilling the statin intolerant definition at moderate CV risk;
* LDL-C ≥160 mg/dL (≥4.1 mmol/L) at screening for participants receiving diet only or, participants not fulfilling the statin intolerant definition at moderate CV risk and receiving a non-statin LMT.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2013-12-16; Primary Completion 2014-10-27 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (43):
- United States (8):
  - Investigational Site Number 840703, Beverly Hills, California
  - Investigational Site Number 840704, Atlantis, Florida
  - Investigational Site Number 840708, Jacksonville, Florida
  - Investigational Site Number 840701, Sarasota, Florida
  - Investigational Site Number 840706, Fall River, Massachusetts
  - Investigational Site Number 840705, St Louis, Missouri
  - Investigational Site Number 840707, Durham, North Carolina
  - Investigational Site Number 840702, Summerville, South Carolina
- Australia (3):
  - Investigational Site Number 036703, Ashford
  - Investigational Site Number 036702, Perth
  - Investigational Site Number 036701, Woolloongabba
- Belgium (3):
  - Investigational Site Number 056702, Antwerp
  - Investigational Site Number 056703, Haine-Saint-Paul
  - Investigational Site Number 056701, Leuven
- Canada (6):
  - Investigational Site Number 124703, Chicoutimi
  - Investigational Site Number 124701, Québec
  - Investigational Site Number 124704, Sherbrooke
  - Investigational Site Number 124706, Toronto
  - Investigational Site Number 124702, Vancouver
  - Investigational Site Number 124705, Victoria
- Denmark (5):
  - Investigational Site Number 208703, Aarhus
  - Investigational Site Number 208702, Esbjerg
  - Investigational Site Number 208701, Glostrup Municipality
  - Investigational Site Number 208704, Hvidovre
  - Investigational Site Number 208705, Køge
- Netherlands (8):
  - Investigational Site Number 528701, Amsterdam
  - Investigational Site Number 528708, Den Helder
  - Investigational Site Number 528702, Hoogeveen
  - Investigational Site Number 528703, Hoorn
  - Investigational Site Number 528706, Rotterdam
  - Investigational Site Number 528709, Sneek
  - Investigational Site Number 528704, Utrecht
  - Investigational Site Number 528707, Venlo
- New Zealand (2):
  - Investigational Site Number 554702, Auckland
  - Investigational Site Number 554701, Christchurch
- Spain (8):
  - Investigational Site Number 724703, A Coruña
  - Investigational Site Number 724707, Barcelona
  - Investigational Site Number 724710, Barcelona
  - Investigational Site Number 724702, Córdoba
  - Investigational Site Number 724705, Granada
  - Investigational Site Number 724709, Sant Joan Despí
  - Investigational Site Number 724706, Santiago de Compostela
  - Investigational Site Number 724701, Zaragoza

REFERENCES:
- [Result] Stroes E, Guyton JR, Lepor N, Civeira F, Gaudet D, Watts GF, Baccara-Dinet MT, Lecorps G, Manvelian G, Farnier M; ODYSSEY CHOICE II Investigators. Efficacy and Safety of Alirocumab 150 mg Every 4 Weeks in Patients With Hypercholesterolemia Not on Statin Therapy: The ODYSSEY CHOICE II Study. J Am Heart Assoc. 2016 Sep 13;5(9):e003421. doi: 10.1161/JAHA.116.003421. PMID 27625344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 43 centers in 8 countries. A total of 402 participants were screened between December-2013 and May-2014, of whom 233 were randomized for double-blind (DB) treatment period and 169 were screen failures. Out of 233 randomized for DB period, 205 participants entered the optional open-label (OL) extension period.
Pre-assignment Details: Randomization was stratified by statin intolerant status & background therapy (non-statin lipid therapy vs diet). Randomization followed a 1:2:1 ratio for placebo, Alirocumab 75 mg and Alirocumab 150 mg instead of 1:1:2 as initially planned due to systematic error in treatment allocation algorithm discovered after all participants were randomized.
Groups:
- Alirocumab 150 mg Q4W/Up to 150 mg Q2W: Period 1: Alirocumab 150 mg SC injection Q4W added to stable non-statin LMT or diet alone for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels at Week 8 were not achieved i.e. LDL-C ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) depending on cardiovascular risk or <30% LDL-C reduction from baseline.
  Period 2: Alirocumab 150 mg SC injection Q4W from Week 24 until second quarter 2017 or until the drug is commercially available in the country, whatever occurred first. Alirocumab dose could be either up-titrated to 150 mg Q2W from Week 36 or maintained according to the investigator judgement and LDL-C values. Subsequent down titration to 150 mg Q4W was allowed.
Period: Period 1: 24-Week Double-blind Treatment
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W (Calibrator) | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Started | 58 | 116 | 59
Treated | 58 | 115 | 58
Completed | 54 | 107 | 50
Not Completed | 4 | 9 | 9
Not completed — Adverse Event | 2 | 2 | 5
Not completed — Poor compliance to protocol | 0 | 2 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Consent withdrawn by participant | 1 | 0 | 1
Not completed — Randomized but not treated | 0 | 1 | 1
Not completed — Other than specified above | 1 | 3 | 1
Period: Extension Open Label Treatment
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W (Calibrator) | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Started | 51 (The open-label extension period was optional for participants who completed the double-blind period.) | 106 (The open-label extension period was optional for participants who completed the double-blind period.) | 48 (The open-label extension period was optional for participants who completed the double-blind period.)
Completed | 46 | 89 | 43
Not Completed | 5 | 17 | 5
Not completed — Adverse Event | 1 | 7 | 3
Not completed — Poor compliance to protocol | 1 | 1 | 0
Not completed — Participant moved | 1 | 2 | 0
Not completed — Other than specified above | 2 | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Alirocumab 150 mg Q4W/Up to 150 mg Q2W: Period 1: Alirocumab 150 mg SC injection Q4W added to stable non-statin LMT or diet alone for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when targeted LDL-C levels at Week 8 were not achieved i.e. LDL-C ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) depending on cardiovascular risk or <30% LDL-C reduction from baseline.
  Period 2: Alirocumab 150 mg SC injection Q4W from Week 24 until second quarter 2017 or until the drug is commercially available in the country, whatever occurred first. Alirocumab dose could be either up-titrated to 150 mg Q2W from Week 36 or maintained according to the investigator judgement and LDL-C values. Subsequent down titration to 150 mg Q4W was allowed.
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W (Calibrator) | Alirocumab 150 mg Q4W/Up to 150 mg Q2W | Total
Number analyzed (Participants) | 58 | 116 | 59 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (10.7) | 62.5 (9.9) | 64.2 (10.0) | 63.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 47 | 29 | 103
  Male | 31 | 69 | 30 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 7 | 4 | 12
  Not Hispanic or Latino | 57 | 109 | 54 | 220
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 4 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 1 | 3 | 1 | 5
  White | 56 | 108 | 55 | 219
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C from Friedewald formula (LDL-C = Total cholesterol [Total-C] - High-Density Lipoprotein Cholesterol [HDL-C] - [Triglyceride/5]).
  mg/dL | 158.5 (47.3) | 154.5 (44.6) | 163.9 (69.1) | 157.9 (52.4)
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] | 4.106 (1.226) | 4.002 (1.154) | 4.245 (1.789) | 4.089 (1.356)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - Intent-to-Treat (ITT Analysis)
Description: Adjusted Least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 24
Population: ITT population that included all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo Q2W: Placebo (for Alirocumab) subcutaneous (SC) injection every 2 weeks (Q2W) added to stable non-statin lipid modifying therapy (LMT) or diet alone for 24 weeks.
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W (Calibrator): Alirocumab 75 mg SC injection Q2W added to stable non-statin LMT or diet alone for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when targeted low-density lipoprotein cholesterol (LDL-C) levels at Week 8 were not achieved i.e. LDL-C ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) depending on cardiovascular risk or <30% LDL-C reduction from baseline.
- Alirocumab 150 mg Q4W/Up to 150 mg Q2W: Alirocumab 150 mg SC injection Q4W added to stable non-statin LMT or diet alone for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when targeted low-density lipoprotein cholesterol (LDL-C) levels at Week 8 were not achieved i.e. LDL-C ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) depending on cardiovascular risk or <30% LDL-C reduction from baseline.
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W (Calibrator) | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percent change | 4.7 (2.3) | -53.5 (1.6) | -51.7 (2.3)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; Alirocumab 150 mg Q4W/up to 150 mg Q2W was compared to placebo group using an appropriate contrast statement; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; Least square (LS) mean difference = -56.4, 95% CI 2-sided [-62.9 to -49.9] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection) (on-treatment analysis).
Time Frame: From Baseline to Week 24
Population: Modified ITT (mITT) population that included all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W: Alirocumab 75 mg SC injection Q2W added to stable non-statin LMT or diet alone for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when targeted low-density lipoprotein cholesterol (LDL-C) levels at Week 8 were not achieved i.e. LDL-C ≥70 mg/dL (1.81 mmol/L) or ≥100 mg/dL (2.59 mmol/L) depending on cardiovascular risk or <30% LDL-C reduction from baseline.
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 56 | 115 | 57
percent change | 5.1 (2.1) | -55.3 (1.5) | -54.6 (2.1)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -59.7, 95% CI 2-sided [-65.6 to -53.8] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM including all available post-baseline data from Week 4 to Week 24 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percent change | 3.2 (2.5) | -50.8 (1.7) | -41.7 (2.4)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -44.9, 95% CI 2-sided [-51.8 to -38.1] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 24
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 56 | 115 | 57
percent change | 3.6 (2.3) | -51.5 (1.6) | -44.8 (2.3)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -48.4, 95% CI 2-sided [-54.8 to -41.9] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

5. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C to Averaged Weeks 9 to 12 - ITT- Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM including all available post-baseline data from Week 4 to Week 24 regardless of status on-or off-treatment and assigning a weight of 0.25 for Week 9, 10, 11 and 12 time points.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percent change | 3.2 (2.0) | -53.6 (1.4) | -52.3 (2.0)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -55.5, 95% CI 2-sided [-61.1 to -49.8] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

6. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Averaged Week 9 to 12 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection) and assigning a weight of 0.25 for Week 9, 10, 11 and 12 time points.
Time Frame: From Baseline to Week 24
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 56 | 115 | 57
percent change | 3.6 (1.9) | -54.1 (1.3) | -55.0 (1.9)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -58.6, 95% CI 2-sided [-63.8 to -53.4] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM including all available post-baseline data from Week 4 to Week 24 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population. Number of participants analyzed = participants of the ITT population with available data at specified time-points.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 56 | 112 | 58
percent change | 7.5 (2.1) | -39.7 (1.5) | -38.9 (2.2)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -46.4, 95% CI 2-sided [-52.4 to -40.4] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

8. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 - On-treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 24
Population: mITT population. Number of participants analyzed = participants of the mITT population with available data at specified time-points.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 54 | 112 | 54
percent change | 7.7 (2.0) | -41.2 (1.4) | -40.9 (2.1)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -48.6, 95% CI 2-sided [-54.3 to -42.8] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

9. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percent change | 4.8 (2.1) | -45.3 (1.5) | -44.2 (2.1)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -49.0, 95% CI 2-sided [-54.9 to -43.2] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

10. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 - On-treatment Analysis
Description: as for outcome 8
Time Frame: From Baseline to Week 24
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 56 | 115 | 57
percent change | 5.0 (1.9) | -46.9 (1.3) | -46.7 (1.9)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -51.7, 95% CI 2-sided [-57.1 to -46.4] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

11. Secondary Outcome: Percent Change From Baseline in Total-C at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percent change | 3.0 (1.6) | -34.0 (1.1) | -32.3 (1.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -35.3, 95% CI 2-sided [-39.8 to -30.8] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

12. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 56 | 112 | 58
percent change | 7.0 (2.2) | -38.4 (1.6) | -31.3 (2.2)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -38.2, 95% CI 2-sided [-44.3 to -32.1] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

13. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percent change | 3.0 (2.2) | -43.4 (1.5) | -34.9 (2.2)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -37.9, 95% CI 2-sided [-43.9 to -31.8] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

14. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percent change | 1.8 (1.6) | -32.6 (1.2) | -24.5 (1.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -26.3, 95% CI 2-sided [-30.9 to -21.7] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

15. Secondary Outcome: Percentage of Very High Cardiovascular (CV) Risk Participants Achieving Calculated LDL-C <70 mg/dL (<1.81 mmol/L) or Moderate or High CV Risk Participants Achieving Calculated LDL-C <100 mg/dL (<2.59 mmol/L) at Week 24 - ITT Analysis
Description: Moderate CV risk: 10-year fatal cardiovascular disease (CVD) risk Systemic Coronary Risk Evaluation (SCORE) ≥1 and <5%.
  High CV risk: 10-year fatal CVD risk SCORE ≥5% or moderate chronic kidney disease or type 1 or type 2 diabetes mellitus without target organ damage or familial hypercholesterolemia.
  Very high CV risk: history of documented coronary heart disease, ischemic stroke, peripheral artery disease, transient ischemic attack, abdominal aortic aneurysm, or carotid artery occlusion >50% without symptoms; carotid endarterectomy or carotid artery stent procedure; renal artery stenosis, or renal artery stent procedure; or type 1 or type 2 diabetes mellitus with target organ damage.
  Adjusted percentages at Week 24 were obtained from a multiple imputation approach model for handling of missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were included.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percentage of participants | 1.8 | 70.3 | 63.9
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 279.8, 95% CI 2-sided [29.1 to 2690.1] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

16. Secondary Outcome: Percentage of Very High CV Risk Participants Achieving Calculated LDL-C< 70 mg/dL (<1.81 mmol/L) or Moderate or High CV Risk Participants Achieving Calculated LDL-C< 100 mg/dL (<2.59 mmol/L) at Week 24 - On-treatment Analysis
Description: Adjusted percentages at Week 24 from multiple imputation approach including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 56 | 115 | 57
percentage of participants | 1.8 | 72.7 | 67.7
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 354.7, 95% CI 2-sided [36.2 to 3479.5] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

17. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C< 70 mg/dL (<1.81 mmol/L) at Week 24 - ITT Analysis
Description: Adjusted percentages at Week 24 from last observation carried forward (LOCF) approach including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percentage of participants | 0.0 | 60.0 | 50.0
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; LOCF approach followed by logistic regression model; Odds Ratio (OR) = 126.0, 95% CI 2-sided [20.0 to 9999] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo (Confidence interval should be read as 20.0 to >9999)

18. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <70 mg/dL (<1.81 mmol/L) at Week 24 - On-treatment Analysis
Description: Adjusted percentages at Week 24 from LOCF approach including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 56 | 115 | 57
percentage of participants | 0.0 | 61.7 | 50.9
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; LOCF approach followed by logistic regression model; Odds Ratio (OR) = 141.5, 95% CI 2-sided [22.2 to 9999] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo (Confidence interval should be read as 20.0 to >9999)

19. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from a multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percent change | 4.1 (3.7) | -21.8 (2.6) | -15.5 (3.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0002, Regression, Robust — Threshold for significance at 0.05 level; Multiple imputation approach followed by robust regression model; Adjusted mean difference = -19.6, 95% CI 2-sided [-29.8 to -9.4] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

20. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 from a multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percent change | 2.2 (3.4) | -16.5 (2.4) | -5.7 (3.3)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 150 mg Q4W/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0892, Regression, Robust — Threshold for significance at 0.05 level; Multiple imputation approach followed by robust regression model; Adjusted mean difference = -7.9, 95% CI 2-sided [-17.1 to 1.2] — Alirocumab 150 mg Q4W/Up to 150 mg Q2W vs. Placebo

21. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percent change | -2.4 (1.9) | 7.4 (1.4) | 7.7 (2.0)

22. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percent change | -0.8 (1.9) | 6.8 (1.3) | 8.6 (1.9)

23. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: as for outcome 19
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percent change | 1.1 (3.8) | -10.6 (2.7) | -9.2 (3.9)

24. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 from a multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 57 | 115 | 58
percent change | 2.1 (3.9) | -11.3 (2.7) | -3.0 (3.8)

25. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 56 | 112 | 58
percent change | 3.4 (1.5) | 8.2 (1.1) | 10.0 (1.5)

26. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 12 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Alirocumab 150 mg Q4W/Up to 150 mg Q2W
Number analyzed (Participants) | 56 | 112 | 58
percent change | 2.6 (1.5) | 5.9 (1.1) | 7.6 (1.5)

27. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 32, 36, 48, 72, 96, 120, 144, 168 On-Treatment Analysis in Open Label Extension Treatment Phase
Description: Mean percent changes (and standard deviations) observed during the open-label extension period are provided.
Time Frame: Baseline, Week 32, 36, 48, 72, 96, 120, 144 and Week 168
Population: Open-label extension population included all participants who received at least one dose or part of dose of Alirocumab during the open label extension period. Here, "number analyzed" signifies the number of participants evaluable for each specified time-point.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Alirocumab 150 mg Q4W (After Placebo Q2W): Alirocumab 150 mg SC injection Q4W from Week 24 until second quarter 2017 or until the drug is commercially available in the country, whatever occurred first, in participants who received placebo (for Alirocumab) Q2W for 24 weeks during the double-blind period. Alirocumab dose could be either up-titrated to 150 mg Q2W from Week 36 or maintained according to the investigator judgement and low-density lipoprotein cholesterol (LDL-C) values. Subsequent down titration to 150 mg Q4W was allowed.
- Alirocumab 150 mg QW4 (After Alirocumab 75 Q2W/Up 150 Q2W): Alirocumab 150 mg SC injection Q4W from Week 24 until second quarter 2017 or until the drug is commercially available in the country, whatever occurred first, in participants who received Alirocumab 75 mg Q2W/Up to 150 mg Q2W for 24 weeks during the double-blind period. Alirocumab dose could be either up-titrated to 150 mg Q2W from Week 36 or maintained according to the investigator judgement and low-density lipoprotein cholesterol (LDL-C) values. Subsequent down titration to 150 mg Q4W was allowed.
- Alirocumab 150 mg Q4W (After Alirocumab 150 Q4W/Up 150 Q2W): Alirocumab 150 mg SC injection Q4W from Week 24 until second quarter 2017 or until the drug is commercially available in the country, whatever occurred first, in participants who received 150 mg Q4W/Up to 150 mg Q2W for 24 weeks during the double-blind period. Alirocumab dose could be either up-titrated to 150 mg Q2W from Week 36 or maintained according to the investigator judgement and low-density lipoprotein cholesterol (LDL-C) values. Subsequent down titration to 150 mg Q4W was allowed.
Arm/Group | Alirocumab 150 mg Q4W (After Placebo Q2W) | Alirocumab 150 mg QW4 (After Alirocumab 75 Q2W/Up 150 Q2W) | Alirocumab 150 mg Q4W (After Alirocumab 150 Q4W/Up 150 Q2W)
Number analyzed (Participants) | 51 | 106 | 48
percent change
  Week 32: number analyzed (Participants) | 48 | 98 | 45
  Week 32 | -37.3 (18.8) | -41.1 (21.2) | -46.9 (13.3)
  Week 36: number analyzed (Participants) | 48 | 96 | 46
  Week 36 | -36.1 (22.0) | -39.2 (21.2) | -43.1 (13.7)
  Week 48: number analyzed (Participants) | 47 | 91 | 44
  Week 48 | -46.5 (24.2) | -49.2 (18.7) | -48.7 (21.7)
  Week 72: number analyzed (Participants) | 50 | 94 | 47
  Week 72 | -50.8 (20.6) | -53.7 (19.5) | -52.3 (21.3)
  Week 96: number analyzed (Participants) | 48 | 90 | 44
  Week 96 | -49.8 (20.4) | -52.8 (19.6) | -46.8 (22.0)
  Week 120: number analyzed (Participants) | 46 | 81 | 37
  Week 120 | -50.6 (20.9) | -53.7 (18.7) | -51.8 (24.1)
  Week 144: number analyzed (Participants) | 38 | 72 | 29
  Week 144 | -52.7 (17.6) | -48.7 (23.7) | -49.4 (20.9)
  Week 168: number analyzed (Participants) | 4 | 13 | 4
  Week 168 | -47.8 (24.2) | -66.2 (17.1) | -60.0 (4.6)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of informed consent form up to study completion (up to 176 weeks) regardless of seriousness or relationship to investigational product.
Description: Reported AEs/deaths are treatment-emergent ie; AEs that developed/worsened and deaths that occurred 'on treatment'; from 1st dose up to last dose (active/placebo depending on Q2W/Q4W dosing) in DB period+70 days, truncated at the day before 1st dose in OL period for participants entering in OL period; from 1st dose up to last dose in OL period+70 days.
Groups:
- Placebo Q2W: Participants exposed to placebo SC injection Q2W added to stable non-statin LMT or diet alone (mean exposure of 23 weeks).
- Alirocumab 75 mg Q2W/Up150 mg Q2W: Participants exposed to alirocumab 75 mg Q2W/up to 150 mg Q2W SC injection added to stable non-statin LMT or diet alone (mean exposure of 23 weeks).
- Alirocumab 150 mg Q4W/Up150 mg Q2W: Participants exposed to alirocumab 150 mg Q4W/up to 150 mg Q2W SC injection added to stable non-statin LMT or diet alone (mean exposure of 22 weeks).
- Alirocumab 150 mg Q4W (After Placebo Q2W): Participants exposed to alirocumab 150 mg Q4W SC injection added to stable non-statin LMT or diet alone (mean exposure of 128 weeks) after having received Placebo Q2W for 24 weeks.
- Alirocumab 150 mg Q4W (After Alirocumab 75 Q2W/Up150 Q2W): Participants exposed to alirocumab 150 mg Q4W SC injection added to stable non-statin LMT or diet alone (mean exposure of 117 weeks) after having received Alirocumab 75 mg Q2W/Up to 150 mg Q2W for 24 weeks.
- Alirocumab 150 mg Q4W (After Alirocumab 150 Q4W/Up150 Q2W): Participants exposed to alirocumab 150 mg Q4W SC injection added to stable non-statin LMT or diet alone (mean exposure of 119 weeks) after having received Alirocumab 150 mg Q4W/Up to 150 mg Q2W for 24 weeks.
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up150 mg Q2W | Alirocumab 150 mg Q4W/Up150 mg Q2W | Alirocumab 150 mg Q4W (After Placebo Q2W) | Alirocumab 150 mg Q4W (After Alirocumab 75 Q2W/Up150 Q2W) | Alirocumab 150 mg Q4W (After Alirocumab 150 Q4W/Up150 Q2W)
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/115 | 0/58 | 0/51 | 2/106 | 1/48
Serious Adverse Events (participants affected / at risk) | 4/58 | 7/115 | 7/58 | 15/51 | 28/106 | 14/48
Other Adverse Events (participants affected / at risk) | 28/58 | 61/115 | 29/58 | 42/51 | 71/106 | 31/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=58) | Alirocumab 75 mg Q2W/Up150 mg Q2W (N=115) | Alirocumab 150 mg Q4W/Up150 mg Q2W (N=58) | Alirocumab 150 mg Q4W (After Placebo Q2W) (N=51) | Alirocumab 150 mg Q4W (After Alirocumab 75 Q2W/Up150 Q2W) (N=106) | Alirocumab 150 mg Q4W (After Alirocumab 150 Q4W/Up150 Q2W) (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 3 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Basedow's disease (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 2 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis E (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Traumatic renal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 2 | 1
Benign fallopian tube neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1 | 2 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Arachnoiditis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=58) | Alirocumab 75 mg Q2W/Up150 mg Q2W (N=115) | Alirocumab 150 mg Q4W/Up150 mg Q2W (N=58) | Alirocumab 150 mg Q4W (After Placebo Q2W) (N=51) | Alirocumab 150 mg Q4W (After Alirocumab 75 Q2W/Up150 Q2W) (N=106) | Alirocumab 150 mg Q4W (After Alirocumab 150 Q4W/Up150 Q2W) (N=48)
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 1 | 3 | 11 | 2
Nausea (Gastrointestinal disorders) | 2 | 6 | 3 | 1 | 3 | 3
Fatigue (General disorders) | 0 | 5 | 4 | 3 | 7 | 3
Injection site reaction (General disorders) | 0 | 4 | 8 | 1 | 7 | 7
Non-cardiac chest pain (General disorders) | 3 | 3 | 0 | 6 | 5 | 1
Oedema peripheral (General disorders) | 4 | 3 | 0 | 4 | 5 | 5
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 3 | 4 | 5
Influenza (Infections and infestations) | 0 | 3 | 1 | 3 | 9 | 4
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 3 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 3 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 3 | 7 | 8 | 4
Urinary tract infection (Infections and infestations) | 1 | 4 | 4 | 4 | 7 | 5
Viral upper respiratory tract infection (Infections and infestations) | 3 | 10 | 5 | 5 | 16 | 9
Fall (Injury, poisoning and procedural complications) | 1 | 6 | 0 | 6 | 14 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 3 | 3 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 5 | 5 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 8 | 7 | 8 | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2 | 4 | 10 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 9 | 3 | 4 | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 1 | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 7 | 3 | 7 | 6 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 8 | 7 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 2 | 3 | 1
Dizziness (Nervous system disorders) | 4 | 1 | 4 | 4 | 5 | 4
Headache (Nervous system disorders) | 4 | 10 | 5 | 3 | 6 | 4
Depression (Psychiatric disorders) | 0 | 2 | 1 | 1 | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 9 | 9 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0 | 3 | 1
Hypertension (Vascular disorders) | 2 | 1 | 2 | 2 | 8 | 2

LIMITATIONS AND CAVEATS:
The systematic randomization error was not anticipated to have an impact on the power of the study. The sample size to detect a difference in efficacy endpoints was reached (it was increased to obtain additional safety data) and blind was maintained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.